CLINICAL TRIAL: NCT05053373
Title: Evaluation of Integrated Optimization Schemes for Female Stress Incontinence
Acronym: EIOSFSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChiCTR-IPR-15006711; 2012BAI24B01 (Other Grant/Funding Number: the Ministry of Science and Technology of PRC)
Record Dates: First submitted 2021-09-21; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Stress Urinary Incontinence in Women
Keywords: Stress Urinary Incontinence; Acupuncture
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A central randomized system of clinical research (provided by the Clinical Evaluation Center of the Chinese Academy of Traditional Chinese Medicine) will be used for randomization. When eligible subjects are enrolled, randomized personnel from each center will log on to the central random online system to apply for a randomized number. Then the participants will be randomly assigned to PFMT+EA group or PFMT+sham EA group at a ratio of 1:1 to one of four hospitals. The following individuals in the trial will be blinded: 1) participants, this will be achieved by using sham EA procedure; (2) Evaluators, evaluation and record of measurements will be conducted by the evaluators who do not know the grouping situation; (3) Statisticians, group allocation will not be revealed until the statistical analyses are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Added to Pelvic Floor Muscle Training (Experimental): Patients will be in a prone position. Bilateral Zhongliao (BL33) and Huiyangacupoint (BL35) will be identified and punctured by an acupuncturist. The electrodes will be placed on the needle handles, and stimulate for 30 minutes at 50 Hz with a current intensity between 1 to 5 mA. PFMT will be performed 3 sets a day (morning, around noon, and night).
  Interventions: Device: Electroacupuncture group; Behavioral: Pelvic floor muscle training
- Sham Electroacupuncture Added to Pelvic Floor Muscle Training (Experimental): The preparation for the patients will be the same as that for the patients who will receive EA. Whereas, instead of using real acupuncture needles, special designed placebo needles (size 0.30 × 25 mm) with the blunt-head will be used in the PFMT+sham EA group to penetrate the fixed pad to the skin surface but without skin penetration. The same procedure for deqi will be performed as in the PFMT+EA group. A special-designed cable (the intermediate wire of the cable is cut off but the appearance is normal) will be used to connect the electrodes to the electroacupuncture machine. Therefore, the electroacupuncture machine appears to work, but does not actually stimulated acupoints. The sham EA treatment will also be maintained for 30 minutes. PFMT will be performed 3 sets a day (morning, around noon, and night),
  Interventions: Device: Sham electroacupuncture group; Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Device: Electroacupuncture group
  Other Names: SDA-V electroacupuncture apparatus(Huatuo,made in China)
  Arms: Electroacupuncture Added to Pelvic Floor Muscle Training
Device: Sham electroacupuncture group
  Other Names: Sham SDZ-V electroacupuncture apparatus(Huatuo,China)
  Arms: Sham Electroacupuncture Added to Pelvic Floor Muscle Training
Behavioral: Pelvic floor muscle training

SUMMARY:
The aim of this study is to determine the effectiveness of PFMT added to EA vs PFMT added sham EA for SUI in women.

DETAILED DESCRIPTION:
We will perform a multicenter, randomized, double-blind, sham-controlled, parallel-group clinical trial in four hospitals in China to compare the effectiveness of EA added to PFMT vs sham EA added to PFMT for women with SUI.

The participated women with SUI will be recruited from four participating hospitals or through community clinics by advertising. Participated hospitals include: Yueyang Hospital of Integrated Traditional Chinese and Western Medicine Affiliated to Shanghai University of Traditional Chinese Medicine (Shanghai, China); Shaanxi Hospital of Traditional Chinese Medicine (Xi'an, China); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Tianjin, China); and Nanjing Hospital of Chinese Medicine Affiliated to Nanjing University of Chinese Medicine (Nanjing, China).

Patients will be screened for eligibility. Chief complaint, medical history, and general characteristics (such as age, race, education level, body mass index, manner of child delivery, menopause) will be obtained. Those who met inclusion criteria and are interested in participating in the study will sign an informed consent form and then make another appointment to complete the baseline data collection, including the 72-hr bladder diary, 1-h pad test, International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score, the weekly mean number of urine pads used). Participants will then be assigned randomly to either a PFMT (3 sets/day for 8 weeks) + EA (3 times per week for 8 weeks) group or a PFMT + sham EA group. The primary and secondary outcome will be measured from week 2 to 32. The participant-reported severity of UI and subjective self-evaluation of therapeutic effects will be recorded. Written informed consent will be obtained from all participants before they are included in the study. All clinical investigations will be conducted according to the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 40-75 years of age
* Involuntary leakage of urine during increased intra-abdominal pressure in the absence of a bladder contraction, such as coughing, sneezing, or other physical activities
* a 1-hour pad test exceeds 1 g
* no other treatments are administered for urinary incontinence currently

Exclusion Criteria:

* Subject has urgency and mixed urinary
* Subjects with pelvic organ prolapse, pregnancy, a history of pelvic surgery, chronic respiratory diseases, urinary tract infection, cardiac pacemaker installation, metal allergy, severe needle fear, and currently taking medications for SUI or psychological disorders.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are 40-75 years of age
Enrollment: 358 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
The change of urine loss | The evaluation will be performed when the participants are first distributed into the groups as a baseline, and then at weeks 2, 4, 6 and 8 of treatment.
  The change of urine loss is measured by the 1-hour urine pad test. The 1-hour pad test will be performed as follows: 1) Empty the bladder and wear a preweighted pad. 2) Drink 500 ml of sodium-free liquid in 15 minutes; 3) walk for half hours, including going up and down stairs; 4) perform the following activity in the remaining 30 minutes: squat and stand up 10 times; cough hard 10 times; run in place for 1 minute; bend down to pick up a small object on the ground 5 times; wash hands for 1 minute with running water. 5) Weigh the pad again to calculate the urine leakage (1 gram equivalent to 1 ml of urine).

SECONDARY OUTCOMES:
The average 24-hour urinary incontinence episodes and reduction of more than 50% | The average 24-hour urinary incontinence episodes and reduction of more than 50% at weeks 2, 4, 6, and 8 of treatment measured by a urinary diary. Reduction more than 50% in urine leakage at week 8 from baseline measured by the 1-hour pad test.
  The average 24-hour urinary incontinence episodes and reduction of more than 50% measured by a urinary diary. Reduction more than 50% in urine leakage at week 8 from baseline measured by the 1-hour pad test.
The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) scores | The evaluation will be performed at baseline, weeks 4, 6, 8 of treatment, and weeks 20 and 32 of follow-up.
  The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) scores (range, 0 [best]-21[worst]), which is recommended by the International Consultation on Urological Diseases (ICUD) to evaluate the frequency and volume of urinary incontinence and its impact on quality of life
Participants using urine pads | week 2-8, week 17-20, week 29-32
  The numbers of participants using urine pads and weekly mean pads usage measured by a urinary diary.
severity of urinary incontinence | weeks 2, 4, 6, and 8
  The participant-reported severity of urinary incontinence at weeks 2, 4, 6, and 8 of treatment (mild leaking, several drops; moderate leaking,wet through underwear; severe leaking, wet through trousers)
Subjective self-evaluation of therapeutic effects | week 2, week 4, week 6, week 8, week 20, week 32
  3 point scoring: totally unhelpful=0, minimally helpful=1, moderately helpful=2, very helpful=3
Incidence of adverse events | the 1-8 weeks
  subcutaneous edema, fatigue, severe pain, palpitations, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuelai Chen, Doctor, Study Chair — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine
Locations (4):
- China (4):
  - Department of Acupuncture and Moxibustion, Nanjing Hospital of Chinese Medicine, Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Department of Acupuncture and Moxibustion, Shaanxi Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi
  - Department of Acupuncture and Moxibustion, Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Acupuncture and Moxibustion, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Data are available for the editorial office and other investigators following reasonable requests. A data use agreement needs to be signed. There may be handling and processing costs, depending on the complexity and scope of the request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year after the data are published
Access Criteria: Data are available for the editorial office and other investigators following reasonable requests. A data use agreement needs to be signed.
URL: http://www.medresman.org.cn/pub/en/proj/projectshow.aspx?proj=1282

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Minassian VA, Bazi T, Stewart WF. Clinical epidemiological insights into urinary incontinence. Int Urogynecol J. 2017 May;28(5):687-696. doi: 10.1007/s00192-017-3314-7. Epub 2017 Mar 20. PMID 28321473
- [Background] Lukacz ES, Santiago-Lastra Y, Albo ME, Brubaker L. Urinary Incontinence in Women: A Review. JAMA. 2017 Oct 24;318(16):1592-1604. doi: 10.1001/jama.2017.12137. PMID 29067433
- [Background] Minassian VA, Stewart WF, Wood GC. Urinary incontinence in women: variation in prevalence estimates and risk factors. Obstet Gynecol. 2008 Feb;111(2 Pt 1):324-31. doi: 10.1097/01.AOG.0000267220.48987.17. PMID 18238969
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Oliveira M, Ferreira M, Azevedo MJ, Firmino-Machado J, Santos PC. Pelvic floor muscle training protocol for stress urinary incontinence in women: A systematic review. Rev Assoc Med Bras (1992). 2017 Jul;63(7):642-650. doi: 10.1590/1806-9282.63.07.642. PMID 28977091
- [Background] Markland AD, Richter HE, Fwu CW, Eggers P, Kusek JW. Prevalence and trends of urinary incontinence in adults in the United States, 2001 to 2008. J Urol. 2011 Aug;186(2):589-93. doi: 10.1016/j.juro.2011.03.114. PMID 21684555
- [Background] Coyne KS, Sexton CC, Thompson CL, Milsom I, Irwin D, Kopp ZS, Chapple CR, Kaplan S, Tubaro A, Aiyer LP, Wein AJ. The prevalence of lower urinary tract symptoms (LUTS) in the USA, the UK and Sweden: results from the Epidemiology of LUTS (EpiLUTS) study. BJU Int. 2009 Aug;104(3):352-60. doi: 10.1111/j.1464-410X.2009.08427.x. Epub 2009 Mar 5. PMID 19281467
- [Background] Waetjen LE, Liao S, Johnson WO, Sampselle CM, Sternfield B, Harlow SD, Gold EB. Factors associated with prevalent and incident urinary incontinence in a cohort of midlife women: a longitudinal analysis of data: study of women's health across the nation. Am J Epidemiol. 2007 Feb 1;165(3):309-18. doi: 10.1093/aje/kwk018. Epub 2006 Nov 28. PMID 17132698
- [Background] Komesu YM, Schrader RM, Ketai LH, Rogers RG, Dunivan GC. Epidemiology of mixed, stress, and urgency urinary incontinence in middle-aged/older women: the importance of incontinence history. Int Urogynecol J. 2016 May;27(5):763-72. doi: 10.1007/s00192-015-2888-1. Epub 2015 Dec 15. PMID 26670573
- [Background] Nambiar AK, Bosch R, Cruz F, Lemack GE, Thiruchelvam N, Tubaro A, Bedretdinova DA, Ambuhl D, Farag F, Lombardo R, Schneider MP, Burkhard FC. EAU Guidelines on Assessment and Nonsurgical Management of Urinary Incontinence. Eur Urol. 2018 Apr;73(4):596-609. doi: 10.1016/j.eururo.2017.12.031. Epub 2018 Feb 3. PMID 29398262
- [Background] KEGEL AH. Progressive resistance exercise in the functional restoration of the perineal muscles. Am J Obstet Gynecol. 1948 Aug;56(2):238-48. doi: 10.1016/0002-9378(48)90266-x. No abstract available. PMID 18877152
- [Background] Qaseem A, Dallas P, Forciea MA, Starkey M, Denberg TD, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Nonsurgical management of urinary incontinence in women: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2014 Sep 16;161(6):429-40. doi: 10.7326/M13-2410. PMID 25222388
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Antonov NM, Lachinova IN. [Ambulatory acupuncture treatment of patients with nocturnal urinary incontinence]. Urol Nefrol (Mosk). 1974;39(4):44-6. No abstract available. Russian. PMID 4408536
- [Background] Kost'al M, Hrubecky I. [Acupuncture in the treatment of female incontinence]. Cesk Gynekol. 1985 Aug;50(7):488-90. No abstract available. Czech. PMID 4042173
- [Background] Kubista E, Altmann P, Kucera H, Rudelstorfer B. Electro-acupuncture's influence on the closure mechanism of the female urethra in incontinence. Am J Chin Med (Gard City N Y). 1976 Summer;4(2):177-81. doi: 10.1142/s0192415x76000226. PMID 945686
- [Background] Xie HZ. [Stress urinary incontinence in the female (analysis of 116 cases (author's transl)]. Zhonghua Fu Chan Ke Za Zhi. 1980;15(2):68-70. No abstract available. Chinese. PMID 7471999
- [Background] Philp T, Shah PJ, Worth PH. Acupuncture in the treatment of bladder instability. Br J Urol. 1988 Jun;61(6):490-3. doi: 10.1111/j.1464-410x.1988.tb05086.x. PMID 3401657
- [Background] Kim JH, Nam D, Park MK, Lee ES, Kim SH. Randomized control trial of hand acupuncture for female stress urinary incontinence. Acupunct Electrother Res. 2008;33(3-4):179-92. doi: 10.3727/036012908803861122. PMID 19301628
- [Background] Wang Y, Zhishun L, Peng W, Zhao J, Liu B. Acupuncture for stress urinary incontinence in adults. Cochrane Database Syst Rev. 2013 Jul 1;2013(7):CD009408. doi: 10.1002/14651858.CD009408.pub2. PMID 23818069
- [Background] Langevin HM, Schnyer R, MacPherson H, Davis R, Harris RE, Napadow V, Wayne PM, Milley RJ, Lao L, Stener-Victorin E, Kong JT, Hammerschlag R; Executive Board of the Society for Acupuncture Research. Manual and electrical needle stimulation in acupuncture research: pitfalls and challenges of heterogeneity. J Altern Complement Med. 2015 Mar;21(3):113-28. doi: 10.1089/acm.2014.0186. Epub 2015 Feb 24. PMID 25710206
- [Background] Abrams P, Khoury S, Cardozo L, Wein A. Incontinence : 5th International Consultation on Incontinence, Paris, February 2012. 2013.
- [Background] Yang XY, Shi GX, Li QQ, Zhang ZH, Xu Q, Liu CZ. Characterization of deqi sensation and acupuncture effect. Evid Based Complement Alternat Med. 2013;2013:319734. doi: 10.1155/2013/319734. Epub 2013 Jun 20. PMID 23864884
- Available data/document: Individual Participant Data Set — http://www.medresman.org.cn/pub/en/proj/projectshow.aspx?proj=1282